CLINICAL TRIAL: NCT00492518
Title: Acetylcysteine, Theophylline, and a Combination of Both in the Prophylaxis of Contrast-Induced Nephropathy: A Placebo Controlled Randomized Study
Brief Title: Acetylcysteine, Theophylline, and a Combination of Both in the Prophylaxis of Contrast-Induced Nephropathy
Acronym: ATHENS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ACC-Theo-1.3
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Last update posted 2007-06-27 (Estimated); Status verified 2007-06

CONDITIONS: Contrast Induced Nephropathy; Kidney Diseases; Renal Failure; Adverse Effects
Keywords: Contrast Induced Nephropathy; Prophylaxis; Theophylline; Acetylcysteine; Coronary angiography
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency | interventions — Acetylcysteine; Theophylline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Acetylcysteine
Drug: Theophylline
Drug: Placebo

SUMMARY:
Several studies demonstrated a significant reduction of contrast-induced nephropathy (CIN; definition: increase in serum creatinine of >=0.5mg/dl and/or >=25% increase within 48h after contrast-medium) by acetylcysteine (A) or theophylline (T). However, the results are contradictory. Therefore, it was the aim of our double-blind study to compare the effects of A, T, a combination of A and T (A+T), and placebo (P).

DETAILED DESCRIPTION:
Contrast-induced nephropathy (CIN) is the third leading cause of hospital-acquired acute renal failure (ARF). Accounting for 12% of ARF cases, CIN is defined as an increase of serum creatinine of at least 0.5 mg/d ("Barrett´s definition") and/or 25% within 48 hours of contrast-medium application. CIN is associated with prolonged hospitalisation and increased mortality. CIN frequency depends on several risk-factors including pre-existing renal dysfunction, high amounts of contrast-medium, diabetes, and concurrent use of nephrotoxic drugs. CIN incidence is low in the absence of risk-factors; however, in high-risk patients, CIN occurs in more than 50% of patients.

A variety of prophylactic approaches have been investigated. Despite nephro-protective effects of hydration with saline or with sodium bicarbonate, other trials reported CIN-incidences between 20 and 50% despite hydration. Several studies and two recent meta-analyses demonstrated a significant reduction of renal impairment after contrast-medium using medical prophylaxis with the adenosine antagonist theophylline. However, a recent trial failed to prove prophylactic effects of theophylline.

The antioxidant acetylcysteine (ACC) was effective in patients with impaired renal function in at least six studies, but it was not preventive in at least 21 trials and two recent meta-analyses. A recent study comparing the prophylactic efficacy of theophylline and acetylcysteine demonstrated superior prophylactic effects of theophylline. Nevertheless, this study did not include a placebo group, was not restricted to patients with impaired renal function and exclusively enrolled ICU-patients.

Therefore, we performed a double-blinded study to compare the effects of acetylcysteine, theophylline, a combination of both, and placebo in patients with impaired renal function (serum creatinine >=1.3mg/dl) parenterally receiving >=100ml of contrast-medium.

ELIGIBILITY:
Inclusion Criteria:

* Impaired renal function (serum creatinine >=1.3mg/dl)
* >=100ml of contrast-medium
* Age >= 18years
* Informed consent

Exclusion Criteria:

* Previous dialysis and/or haemofiltration
* Pre-treatment with acetylcysteine and/or theophylline within the last 2 days,
* Pregnancy
* Contraindications to theophylline (untreated high grade arrhythmia or a history of seizures) or acetylcysteine (known allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2002-02; Study Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
The incidence of contrast induced nephropathy, defined as an increase of serum creatinine of at least 0.5 mg/d and/or 25% within 48 hours of contrast-medium application (comparison of treatment groups to placebo) | 48h after the application of contrast-medium

SECONDARY OUTCOMES:
Change in serum creatinine 48h after contrast medium compared to pre-contrast serum creatinine. Multiple regression analysis of risk-factors of CIN with "Y=Maximum increase of serum creatinine compared to baseline within 48h" | 48h

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Huber, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinikum Rechts der Isar; Technical University of Munich, Munich, Germany